CLINICAL TRIAL: NCT00379548
Title: A Pilot Study of the Changes in Inflammatory State in Asian Americans Changing From Traditional Asian Diet to Typical American Diets
Brief Title: Changes in Inflammatory State in Asian Americans Changing From Traditional Asian Diets to American Diet - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Sunstar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 04-47
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Insulin Resistance; Inflammation; Cardiovascular Disease; Periodontal Disease
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Inflammation; Cardiovascular Diseases; Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Control group- subjects are on the Asian diet for the entire duration of the study
- 2 (Experimental): Asian and Caucasian subjects switch from an Asian Diet to a Western Diet midway through the study.
  Interventions: Behavioral: 2 groups of population responding to 2 types of diets

INTERVENTIONS:
Behavioral: 2 groups of population responding to 2 types of diets — Intervention groups include: Asian intervention and Caucasian intervention- both these groups switch from an Asian diet to a Western diet halfway through the study.
  Arms: 2

SUMMARY:
We hypothesize that Asian Americans compared to Caucasians, will be at higher risk of developing a pro-inflammatory state that may contribute to the development of heart disease and diabetes when they change from a traditional Asian diet to a typical Western diet. These inflammatory responses will be reflected by the activation of monocytes as measured by protein kinase C (PKC), a known activator of monocytes.

We also hypothesize that the changes of these inflammatory responses in the gingival crevicular fluid (GCF) will reflect similar changes of these markers in the plasma and monocytes.

Specific aims:

1. To compare the inflammatory responses (primarily PKC activation in monocytes), between Far-East Asian Americans and Caucasian Americans, when they change from a traditional Asian diet to a typical American diet.
2. To correlate the biochemical changes of inflammatory responses in the plasma and monocytes with those in the gingival crevicular fluid (GCF).

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian or Far-East Asian decent
2. Ages between 25 - 55 years old
3. Has family history of diabetes defined as having a first degree relative diagnosed with diabetes mellitus, and/or medical history of gestational diabetes (GDM), impaired fasting glucose(IFG) and impaired glucose tolerance (IGT)
4. BMI of 18.5 - 25.0 kg/m2
5. Agree to maintain constant physical activity levels for the duration of the study
6. Agree to utilize contraception for the duration of the study (for female subjects)
7. Have a minimum of 12 natural teeth
8. Scoring of 2 or more on dental screening questionnaire (See appendix)
9. Ability to communicate in English

Exclusion Criteria:

1. Acute weight loss/weight gain over the past 6 months (defined as +4 lbs or more/month)
2. History of diabetes
3. Current Smokers (including those who quit < 1 year)
4. Heavy alcohol drinkers, defined as drinking more than 7 drinks/week. Those who drink alcohol will need to be reported and documented. They will be asked to maintain the levels of alcohol consumption throughout the study.
5. Medical history of vascular diseases (CAD, MI, stroke, CABG, angioplasty), diabetes, liver disease, kidney disease, cancer, AIDS, bleeding disorders
6. History of food allergies or to any food products in the diet menu.
7. Enrolled in another investigational study within 1 month prior to screening for this study
8. Vegetarian, those with significant food aversions, and anyone who cannot comply with the diet
9. Pregnancy or breasting feeding
10. Other autoimmune or inflammatory conditions or diseases that may compromise the patient's safety or compliance during the study on an individual basis
11. Chronic use of antibiotics or anti-inflammatory medications (>1 month) within the past year
12. On medications such as statins, angiotensin converting enzyme inhibitor, warfarin, aspirin or other anti-inflammatory medications. Daily multivitamins are permitted, excluding pharmacological doses of anti- oxidants will not be allowed.
13. Individuals with dental needs requiring extensive dental restorations such as cavities, root canals, crowns, etc.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in inflammatory markers including PKC and IL6 and Gingival Crevicular Fluid | before Asian Diet, after 8 weeks of Asian Diet, after 8 weeks of Western Diet
Lipid profiles | before Asian Diet, after 8 weeks of Asian Diet, after 8 weeks of Western Diet
Blood glucose levels | before Asian Diet, after 8 weeks of Asian Diet, after 8 weeks of Western Diet
Body Fat percentage assessed by Dual X-ray Absorption | before Asian Diet, after 8 weeks of Asian Diet, after 8 weeks of Western Diet
Insulin resistance assessed by HOMA | before Asian Diet, after 8 weeks of Asian Diet, after 8 weeks of Western Diet

CONTACTS AND LOCATIONS:
Overall Officials: George L King, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hsu WC, Lau KH, Matsumoto M, Moghazy D, Keenan H, King GL. Improvement of insulin sensitivity by isoenergy high carbohydrate traditional Asian diet: a randomized controlled pilot feasibility study. PLoS One. 2014 Sep 16;9(9):e106851. doi: 10.1371/journal.pone.0106851. eCollection 2014. PMID 25226279